CLINICAL TRIAL: NCT02557035
Title: A Phase 3, Single-dose, Multicenter, Randomized, Double-blind, Parallel Group Study to Assess the Efficacy and Safety of Palonosetron 0.25 mg Administered as a 30-minute IV Infusion Compared to Palonosetron 0.25 mg Administered as a 30-second IV Bolus for the Prevention of Chemotherapy-induced Nausea and Vomiting in Cancer Patients Receiving Highly Emetogenic Chemotherapy.
Brief Title: An Efficacy and Safety Study of Intravenous Palonosetron Administered as an Infusion and as a Bolus for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALO-15-17
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I.V. palonosetron infusion plus dexamethasone (Experimental): Intravenous palonosetron (Aloxi 0.25 mg solution for injection) as an infusion with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Interventions: Drug: Palonosetron; Drug: Dexamethasone
- I.V. palonosetron bolus plus dexamethasone (Active Comparator): Intravenous palonosetron (Aloxi 0.25 mg solution for injection) as a bolus with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Interventions: Drug: Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Palonosetron
Drug: Dexamethasone

SUMMARY:
PALO-15-17 is a clinical study assessing efficacy and safety of a single dose of palonosetron 0.25 mg administered as a 30-minute IV infusion compared to palonosetron 0.25 mg administered as a 30-second IV bolus (Aloxi, an antiemetic drug), both given with oral dexamethasone. The objective of the study is to demonstrate that infused IV palonosetron 0.25 mg is as effective as (non-inferior to) injected palonosetron IV 0.25 mg to prevent nausea and vomiting induced by highly emetogenic cancer chemotherapy in the 0-24 hours after administration of a single cycle of highly emetogenic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically confirmed solid tumor malignancy.
* Naïve to cytotoxic chemotherapy. Previous biological or hormonal therapy will be permitted.
* Scheduled to receive first course of one of the following reference HEC, alone or in combination with other chemotherapeutic agents on Day 1:

  * cisplatin administered as a single IV dose of ≥ 70 mg/m2
  * cyclophosphamide ≥1500 mg/m2
  * carmustine (BCNU) >250 mg/m2
  * dacarbazine (DTIC)
  * mechloretamine (nitrogen mustard)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2 .
* If a patient is female, she shall be of non-childbearing potential or of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test.
* Hematologic and metabolic status adequate for receiving an highly emetogenic regimen based on laboratory criteria (Total Neutrophils,Platelets, Bilirubin, Liver enzymes, Serum Creatinine or Creatinine Clearance)
* Able to read, understand, follow the study procedure and complete patient diary.

Exclusion Criteria:

* Lactating woman.
* Current use of illicit drugs or current evidence of alcohol abuse.
* Scheduled to receive moderately emetogenic chemotherapy or highly emetogenic chemotherapy from Day 2 to Day 5.
* Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to the start of the reference HEC administration on Day 1 or between Days 1 to 5.
* Any vomiting, retching, or nausea (grade ≥ 1 as defined by National Cancer Institute) within 24 hours prior to the start of the reference HEC administration on Day 1.
* Symptomatic primary or metastatic CNS malignancy.
* Active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, an active infection or any illness or medical conditions (other than malignancy) that, in the opinion of the Investigator, may confound the results of the study, represent another potential etiology for emesis and nausea (other than chemotherapy-induced nausea and vomiting) or pose unwarranted risks in administering the study drugs to the patient.
* Known hypersensitivity or contraindication to 5-HT3 receptor antagonists
* Known contraindication to the IV administration of 50 mL 5% glucose solution.
* Participation in a previous clinical trial involving palonosetron.
* Any investigational drugs (other than those given in this study) taken within 4 weeks prior to Day 1, and/or is scheduled to receive any investigational drug during the present study.
* Systemic corticosteroid therapy at any dose within 72 hours prior to the start of the reference HEC administration on Day 1. However, topical and inhaled corticosteroids are permitted.
* Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy.
* Any medication with known or potential antiemetic activity within 24 hours prior to the start of the reference HEC administration on Day 1, including but not limited to 5-HT3 receptor antagonists and NK-1 receptor antagonists
* Concurrent medical condition that would preclude administration of dexamethasone for 4 days such as systemic fungal infection or uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (76):
- Belarus (2):
  - N.N. Aleksandrov Republican Research Oncology and Medical Radiology Center, Department of Chemotherapy, Lesnoy
  - Minsk City Clinical Oncology Center, Minsk
- University Clinical Centre of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment, Dobrich, Department of Medical Oncology, Dobrich
  - Specialized Hospital for Active Treatment in Oncology, Haskovo, Department of Medical Oncology, Haskovo
  - Multiprofile Hospital for Active Treatment "Central Onco Hospital", Plovdiv, Department of Medical Oncology, Plovdiv
  - Complex Oncology Center, Ruse, Department of Medical Oncology, Rousse
  - Multiprofile Hospital for Active Treatment "Serdika", Sofia, Department of Medical Oncology, Sofia
  - University Multiprofile Hospital for Active Treatment "Sveti Ivan Rilski", Sofia, Department of Medical Oncology, Sofia
  - Multiprofile Hospital for Active Treatment for Wonen's Health "Nadezhda", Sofia
  - Hospital for Active Treatment of Oncological Diseases "Dr. Marko Antonov Markov", Varna, Department of Medicinal Oncology and Palliative Care, Varna
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Varna, Clinic of Medical Oncology, Varna
- Georgia (4):
  - JSC NeoMedi, Tbilisi
  - LTD Institute of Clinical Oncology, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LDT High Technology Medical Center University Clinic, Tbilisi
- Greece (4):
  - "Sotiria" Chest Diseases Hospital of Athens, Athens
  - Thermi Clinic S.A., Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", University Department of Pulmonology, Thessaloniki
  - Bioclinic Thessalonikis S.A., Thessaloniki
- Hungary (8):
  - Koranyi National Institute of TBC and Pulmonology, Budapest
  - Uzsoki Hospital, Department of Radiation Oncology, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Petz Aladar County Teaching Hospital, Center for Oncoradiology, Győr
  - Kaposi Mor Teaching Hospital, Centre for Clinical Oncology, Kaposvár
  - Borsod-Abauj-Zemplen County Hospital and University Educational Hospital, Miskolc
  - Szabolcs-Szatmar-Bereg County Hospitals and University Teaching Hospital, Nyíregyháza
  - Medical Center of the University of Pecs, Pécs
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Oncology Hospital, Department of Conservative Oncology, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Clinic of Oncology and Hematology, Kaunas
- Romania (12):
  - Oncopremium Team SRL, Department of Oncology, Baia Mare
  - Prof. Dr. Alexandru Trestioreanu Institute of Oncology, Medical Oncology Department II, Bucharest
  - Coltea Clinical Hospital, Department of Medical Oncology, Bucharest
  - Hifu Terramed Conformal SRL, Department of Medical Oncology, Bucharest
  - Ianuli Med Consult SRL, Oncology Department, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Radiotherapy Department I, Cluj-Napoca
  - Radiotherapy Center Cluj SRL, Department of Oncology, Cluj-Napoca
  - Constanta Emergency Clinical County Hospital, Department of Medical Oncology, Constanța
  - Oncology Center "Sf. Nectarie", Department of Medical Oncology, Craiova
  - Suceava Sf. Ioan cel Nou Emergency County Hospital, Department of Medical Oncology, Suceava
  - Oncomed SRL, Department of Medical Oncology, Timișoara
  - Oncocenter Clinical Oncology SRL, Department of Medical Oncology, Timișoara
- Russia (34):
  - Arkhangelsk Clinical Oncology Center, Arkhangelsk
  - Altay Territorial Oncology Center, Barnaul
  - Bryansk Regional Oncology Center, Bryansk
  - Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - Evimed, LLC, Chelyabinsk
  - Ivanovo Regional Oncology Center, Ivanovo
  - Kaluga Regional Oncology Center, Kaluga
  - Republican Clinical Oncology Center, Kazan'
  - Krasnoyarsk A.I. Kryzhanovsky Regional Oncology Center, Krasnoyarsk
  - Moscow City Oncology Hospital #62, Moscow
  - Moscow Clinical Scientific and Practical Center, Moscow
  - N.N. Blokhin Russian Oncology Research Center, Surgery Dept. 2, Moscow
  - N.N. Blokhin Russian Oncology Research Center, Surgery Dept. of Female Reproductive System Tumors, Moscow
  - N.N. Blokhin Russian Oncology Research Center, Moscow
  - Branch #1 of Nizhny Novgorod Regional Oncology Center, Nizhny Novgorod
  - City Clinical Hospital #1, Novosibirsk
  - Novosibirsk Regional Oncology Center, Novosibirsk
  - Clinical Oncology Center, Dept. of Chemotherapy, Omsk
  - Clinical Oncology Center, Omsk
  - Orenburg Regional Clinical Oncology Center, Orenburg
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Regional Clinical Oncology Center, Ryazan
  - City Clinical Oncology Center, Thoracic Oncology Dept., Saint Petersburg
  - City Clinical Oncology Center, Urology Oncology Dept., Saint Petersburg
  - City Clinical Oncology Center, Saint Petersburg
  - First I.P. Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - St.Petersburg Municipal Clinical Oncology Center, Saint Petersburg
  - Samara Regional Clinical Oncology Center, Samara
  - Tambov Regional Oncology Center, Tambov
  - Tomsk Research Institute of Oncology, General Oncology Dept., Tomsk
  - Tomsk Research Institute of Oncology, Tomsk
  - Republican Clinical Oncology Center, Ufa
  - Regional Clinical Oncology Center, Veliky Novgorod
  - Sverdlovsk Regional Oncology Center, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- I.V. Palonosetron Infusion Plus Dexamethasone: Intravenous palonosetron (Aloxi 0.25 mg solution for injection) as an infusion with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Palonosetron
  Dexamethasone
- I.V. Palonosetron Bolus Plus Dexamethasone: Intravenous palonosetron (Aloxi 0.25 mg solution for injection) as a bolus with oral dexamethasone, both given on Day 1, prior to the scheduled start of cisplatin; then dexamethasone from Days 2 through 4.
  Palonosetron
  Dexamethasone
Period: Overall Study
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Started | 225 | 215
Completed | 218 | 206
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone | Total
Number analyzed (Participants) | 225 | 215 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (8.7) | 58.9 (8.5) | 59.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 71 | 145
  Male | 151 | 144 | 295
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 225 | 215 | 440
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Scale is a standard criteria for measuring how the cancer disease impacts a patient's daily living abilities (known to physicians and researchers as a patient's performance status). It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). There 6 grades, where the performance gets worsening from 0 (patient is fully active, able to carry on all pre-disease performance without restriction) to 5 (patient is dead).
  Participants
    Grade 0 | 97 | 109 | 206
    Grade 1 | 120 | 100 | 220
    Grade 2 | 8 | 6 | 14
Alcohol consumption [Count of Participants; unit: Participants]
  None | 160 | 145 | 305
  Occasional | 58 | 67 | 125
  Regular | 7 | 3 | 10
Tobacco consumption [Count of Participants; unit: Participants]
  non-smoker | 81 | 77 | 158
  Ex-smoker | 81 | 70 | 151
  Regular | 60 | 66 | 126
  Occasional | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 186 | 186

2. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 170 | 165

3. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 150 | 156

4. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 186 | 190

5. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 176 | 168

6. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 155 | 160

7. Secondary Outcome: Percentage of Patients With no Rescue Medication in the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 200 | 195

8. Secondary Outcome: Percentage of Patients With no Rescue Medication in the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 183 | 176

9. Secondary Outcome: Percentage of Patients With no Rescue Medication in the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
Number analyzed (Participants) | 225 | 215
Participants | 173 | 169

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | I.V. Palonosetron Infusion Plus Dexamethasone | I.V. Palonosetron Bolus Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/225 | 0/215
Serious Adverse Events (participants affected / at risk) | 15/225 | 12/215
Other Adverse Events (participants affected / at risk) | 14/225 | 22/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | I.V. Palonosetron Infusion Plus Dexamethasone (N=225) | I.V. Palonosetron Bolus Plus Dexamethasone (N=215)
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 1
Death (General disorders) | 0 | 2
Disease progression (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
ECG signs of myocardial infarction (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | I.V. Palonosetron Infusion Plus Dexamethasone (N=225) | I.V. Palonosetron Bolus Plus Dexamethasone (N=215)
Neutropenia (Blood and lymphatic system disorders) | 8 | 11
Asthenia (General disorders) | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less